CLINICAL TRIAL: NCT00198172
Title: Phase II Study of Cisplatin Plus Epirubicin Salvage Chemotherapy in Refractory Germ Cell Tumors
Brief Title: Phase II Study of Cisplatin Plus Epirubicin Salvage Chemo in Refractory Germ Cell Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual Goal Met
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Indiana University (Other)
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0008-02
Record Dates: First submitted 2005-09-08; First posted 2005-09-20 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Germ Cell Tumor
Keywords: Germ Cell Tumor; Refractory Germ Cell Tumors; Cisplatin plus Epirubicin Salvage Chemotherapy
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Cisplatin; Epirubicin

INTERVENTIONS:
Drug: Cisplatin plus Epirubicin

SUMMARY:
This study proposes to evaluate the combination of cisplatin plus epirubicin in patients with refractory germ cell tumor not amendable to cure with surgery or standard platinum salvage chemotherapy. This regimen will be used in eligible patients after progression on ECOG Study E39897.

DETAILED DESCRIPTION:
To determine the feasibility and toxicity of combining epirubicin to fixed does cisplatin; to determine the partial and complete response rate and duration of remission; to determine the toxicity; to ascertain the potential for greater than 12 month continuous disease-free survival and, therefore, potential curability.

ELIGIBILITY:
Inclusion Criteria:

* histologic or serologic proof of metastatic germ cell neoplasm(gonadal or extragonadal primary) w/ disease not amenable to cure with either surgery or chemotherapy. Pts w/ seminoma & non-seminoma are eligible, as are women w/ ovarian germ cell tumors.
* Must have failed initial cisplatin combination therapy administered w/ curative intent. In addition, pts should have failed and demonstrated progressive disease following the administration of at least one "salvage" regimen for advanced germ cell neoplasms unless they have primary mediastinal nonseminomatous germ cell tumor, or are considered to be a late relapse (>2 yrs since becoming a complete response).
* Pts must have adequate system function (WBC>/= 4,000 & plts >/=100,000; SGOT </=4x normal; bilirubin </=2.0; serum crt </=2.5) obtained </= 4 wks prior to entry.
* ECOG performance status of 0,1, or 2.
* Pts must be at least 3 weeks post major surgery, radiotherapy, or chemotherapy, and have recovered from all toxicity.
* Exclusion Criteria:
* Active, unresolved infection and/or are receiving concurrent treatment w/ parenteral antibiotics. *Eligible after antibiotics have been discontinued for at least 7 days.
* Pregnant or lactating
* Progression w/in 4 wks of lst course of cisplatin combination chemotherapy.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37
Dates: Start 2000-10; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility and toxicity of combining epirubicin to fixed dose cisplatin

SECONDARY OUTCOMES:
To determine the partial and complete response rate and duration of remission

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Einhorn, M.D., Principal Investigator — Indiana University
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States